CLINICAL TRIAL: NCT04408365
Title: Endothelial Function, Inflammation, and Organ Dysfunction in Critically Ill Patients With COVID-19
Brief Title: Endothelial Function, Inflammation and Organ Dysfunction in COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 282930
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: COVID; Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Daily blood samples from ICU admission until day 7 and around the onset of vasodilatory shock Daily urine and RRT effluent fluid samples (if available) from ICU admission until day 7
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients: Adult COVID-19 patients admitted to intensive care units

SUMMARY:
COVID-19 is a rapidly evolving pandemic with approximately 5% of all patients which require intensive care unit admission. In critically ill patients infected with COVID-19, approximately 15% had severe shock requiring medications to increase blood pressure. It appears that blood vessel tone is altered and microcirculation is not well regulated in patients with COVID-19. The underlying pathophysiology and contributing factors are unknown. The association with subsequent organ dysfunction and outcome is also unclear. Therefore, the investigators aim to investigate serial changes of relevant biomarkers in this population to improve the understanding of this disease, to investigate the association with clinically important outcomes and to find out how best to treat patients. The data will serve to develop strategies for individualised management of this high-risk group.

DETAILED DESCRIPTION:
COVID-19 is a rapidly evolving pandemic with approximately 5% of all patients requiring admission to an intensive care unit. In critically ill patients infected with COVID-19, acute respiratory distress syndrome (ARDS) is found in 40%, 11.9% required continuous renal replacement therapy (RRT), and 13.4% had vasodilatory shock.

Currently, supportive treatment is the mainstay treatment, with fluid administration and vasopressors for haemodynamic support and lung-protective ventilation in patients with severe respiratory failure.3 Targeted drugs, antiviral therapies, and vaccines are still currently being developed, but there is currently insufficient evidence to recommend any drug over another.

Dysregulation of vasomotor tone and alteration of microcirculatory function are common in patients infected with COVID-19. The underlying pathophysiology and contributing factors are unknown. The association with subsequent organ dysfunction and outcome is also unclear.

Circulating bio-adrenomedullin regulates vascular tone and endothelial permeability during sepsis, and has been shown to associate with 28-day mortality, vasopressor requirement, RRT, and positive fluid balance. Proenkephalin is a biomarker of glomerular function, and was shown to elevate in patients with acute kidney injury (AKI), especially in those with persistent AKI, and major adverse kidney events. Dipeptidyl peptidase 3 (DPP-3) is a myocardial depressant factor, which is involved in angiotensin II cleavage. High DPP-3 levels were associated with severe organ dysfunction and short-term mortality. In critically ill patients, COVID-19 has been reported to be associated with cardiovascular dysfunction and high mortality.

The renin-angiotensin-aldosterone system (RAAS) may be linked to the pathogenesis of COVID-19. The coronavirus receptor utilizes angiotensin converting enzyme 2 (ACE2) to enter target cells. Endogenous angiotensin II is hypothesized to prevent binding of coronavirus to ACE2, causing internalization and downregulation of ACE2, and causing lysosome-mediated destruction of ACE2. There are no human studies in COVID-19 patients to confirm this hypothesis yet.

There is very little knowledge of underlying pathogenesis in patients with COVID-19 and vasodilatory shock. Therefore, the investigators aim to investigate serial changes of relevant biomarkers in this population to give further understanding of this disease and to investigate the association with clinically important outcomes. The data will serve to develop strategies for individualized management of this high-risk group.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old) admitted to intensive care units
2. Confirmed or suspected severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) infection resulting in coronavirus disease 2019 (COVID-19)

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult COVID-19 patients who are admitted in intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of plasma bio-adrenomedullin | Day 1-7 after intensive care unit admission
  Change of plasma bio-adrenomedullin
Change of plasma proenkephalin | Day 1-7 after intensive care unit admission
  Change of plasma proenkephalin
Change of plasma dipeptidyl peptidase-3 | Day 1-7 after intensive care unit admission
  Change of plasma dipeptidyl peptidase-3
Change of plasma renin | Day 1-7 after intensive care unit admission
  Change of plasma renin
Change of plasma angiotensin II | Day 1-7 after intensive care unit admission
  Change of plasma angiotensin II

SECONDARY OUTCOMES:
Duration of vasodilatory shock | 7 and 28 days
  Duration of vasodilatory shock
Acute kidney injury | 7 and 28 days
  As defined by the Kidney Disease: Improving Global Outcomes criteria
Need for renal replacement therapy | 7 and 28 days
  Need for renal replacement therapy
Duration of ventilation | 7 and 28 days
  Duration of ventilation
Duration of extracorporeal membrane oxygenation | 7 and 28 days
  Duration of extracorporeal membrane oxygenation
Mortality | 28 days
  ICU and hospital

CONTACTS AND LOCATIONS:
Overall Officials: Nuttha Lumlertgul, MD, PhD, Principal Investigator — Guy's & St Thomas' Hospital
Locations (1):
- Guy's & St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided